CLINICAL TRIAL: NCT04105400
Title: Role of Procalcitonin as an Early Marker in Diagnosis of Sepsis in Critically Ill Patient
Brief Title: Procalcitonin in Diagnosis of Sepsis in Critically Ill Patient
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelnasser Mahmoud Ali, resident doctor, Assiut University
Other Study IDs: PCT value in sepsis
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Sepsis, Severe
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
correlation between procalcitonin levels and the severity of sepsis and it's possibility to be used as a prognostic marker in patients with sepsis and severe sepsis

DETAILED DESCRIPTION:
Sepsis is the systemic response to infection by microbial organisms and is considered the leading cause of mortality in patients admitted to intensive care units (ICUs). Audits of ICU worldwide showed that 29.5% patients had sepsis on admission or during the ICU stay The signs and symptoms of sepsis are highly variable and are influenced by many factors, including the virulence and bioburden of the pathogen, the portal of entry, and the host susceptibility.

Early diagnosis of sepsis is often difficult in clinical practice, whilst it can be vital for positive patient outcomes in sepsis management. Any delay in diagnosis and treatment may lead to significant organ failure and can be associated with elevated mortality rates.

Rapid effective management of sepsis not only allows for prompt antibiotic therapy and a potential reduction in mortality, it can also minimize the unnecessary use of antibiotics.

Historically, blood cultures have been the gold standard for diagnosing sepsis, however the lenthy time to generate results is a limitation. Additionally, many patients may have already been prescribed antibiotics prior to arrival to the hospital, which may mask the presentation of sepsis in the blood culture. Despite an emphasis on isolating a specific micro organism, on average, only 34% of blood cultures are found to be positive in septic patients Therefore, while it can be useful, relying on the bacteriological diagnosis can be misleading or too late. A number of the inflammatory markers, such as leukocyte cell count, C reactive protein (CRP), and cytokines (TNF-α, IL-1β, or IL-6), have been applied in the diagnosis of inflammation and infection, but their lack of specificity has generated a continued interest to develop more specific clinical laboratory tests One promising marker has been procalcitonin (PCT), whose concentration has been found to be elevated in sepsis. Owing its specificity to bacterial infections, PCT has been proposed as a pertinent marker in the rapid diagnosis of bacterial infection, especially for use in hospital emergency departments and intensive care units.

PCT has been used as marker of sepsis with sensitivity and specificity of 83% and 62% respectively with significantly high levels in the patients having sepsis and positive blood culture results than with culture negative results PCT is a glycoprotein present in C cells of thyroid gland. It belongs to the group of related peptide (C-GRP) encoded by the CALC-1 gene and is formed from the common precursor pre-calcitonin. In healthy subjects, CALC-1 genes synthesize calcitonin, but presence of microbial infection through endotoxin or proinflammatory cytokines increases calcitonin gene expression and PCT mRNA is mostly synthesized. This lead to release of PCT from all parenchymal tissue, exclusively in response to bacterial infection only and not viral or inflammatory disease Previous studies have demonstrated that procalcitonin levels are correlated with the severity of sepsis and could potentially be used as a prognostic marker in patients with sepsis and severe sepsis In this study we evaluated the usefulness of procalcitonin as a diagnostic predictive marker of bacteremia and sepsis in critically ill patients. Serum PCT levels area useful diagnostic tool available to physicians that can help as a marker of sepsis, as well as other bacterial infections. Combination of emerging new biomarkers with PCT could be used in terms of good clinical judgement based on which antimicrobial therapy may suggested, thus reducing the prescription and duration of antibiotic treatment .

ELIGIBILITY:
Inclusion Criteria:

* adult patients >18 years who were admitted to intensive care unit of Assiut University Hospital with symptoms of systemic infection and with a clinical suspicion of sepsis as guided by the ICU physician

Exclusion Criteria:

* Patients above 70 years of age
* Patients who received antibiotic therapy within three days prior to sample collection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients will be subjected to:
  * Full history & clinical examination.
  * Routine laboratory investigations including:
    * Complete blood count (CBC), with special attention to white blood cells (number & diff.)
    * Serum C-reactive protein (CRP) level
    * Erythrocyte sedimentation rate (ESR)
  Special investigations:
  ● Blood culture : Blood culture will be processed using the Bact/Alert continuous blood culture monitoring system. Bacteria from positive blood cultures will further identified using standard laboratory methods.
  Cultures that did not indicate growth within 5 days of incubation will be considered negative.
  ● Serum procalcitonin will be estimated by ELISA kit.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
role of procalcitonin in early diagnosis of sepsis | Baseline
  Descriptive cross sectional study would be conducted on adult patients >18 years who were admitted to intensive care unit of Assiut University Hospital with symptoms of systemic infection and with a clinical suspicion of sepsis as guided by the ICU physician

REFERENCES:
- [Background] Granic M, Zdravkovic D, Krstajic S, Kostic S, Simic A, Sarac M, Ivanovic N, Radovanovic D, Dikic S, Kovcin V. Totally implantable central venous catheters of the port-a-cath type: complications due to its use in the treatment of cancer patients. J BUON. 2014 Jul-Sep;19(3):842-6. PMID 25261677
- [Background] Vincent JL, Marshall JC, Namendys-Silva SA, Francois B, Martin-Loeches I, Lipman J, Reinhart K, Antonelli M, Pickkers P, Njimi H, Jimenez E, Sakr Y; ICON investigators. Assessment of the worldwide burden of critical illness: the intensive care over nations (ICON) audit. Lancet Respir Med. 2014 May;2(5):380-6. doi: 10.1016/S2213-2600(14)70061-X. Epub 2014 Apr 14. PMID 24740011
- [Background] Karlsson S, Heikkinen M, Pettila V, Alila S, Vaisanen S, Pulkki K, Kolho E, Ruokonen E; Finnsepsis Study Group. Predictive value of procalcitonin decrease in patients with severe sepsis: a prospective observational study. Crit Care. 2010;14(6):R205. doi: 10.1186/cc9327. Epub 2010 Nov 15. PMID 21078153
- [Background] Ruiz-Alvarez MJ, Garcia-Valdecasas S, De Pablo R, Sanchez Garcia M, Coca C, Groeneveld TW, Roos A, Daha MR, Arribas I. Diagnostic efficacy and prognostic value of serum procalcitonin concentration in patients with suspected sepsis. J Intensive Care Med. 2009 Jan-Feb;24(1):63-71. doi: 10.1177/0885066608327095. Epub 2008 Dec 2. PMID 19054806
- [Background] Kim JH, Seo JW, Mok JH, Kim MH, Cho WH, Lee K, Kim KU, Jeon D, Park HK, Kim YS, Kim HH, Lee MK. Usefulness of plasma procalcitonin to predict severity in elderly patients with community-acquired pneumonia. Tuberc Respir Dis (Seoul). 2013 May;74(5):207-14. doi: 10.4046/trd.2013.74.5.207. Epub 2013 May 31. PMID 23750168
- [Background] Novotny A, Emmanuel K, Matevossian E, Kriner M, Ulm K, Bartels H, Holzmann B, Weighardt H, Siewert JR. Use of procalcitonin for early prediction of lethal outcome of postoperative sepsis. Am J Surg. 2007 Jul;194(1):35-9. doi: 10.1016/j.amjsurg.2006.10.026. PMID 17560906
- [Background] Lee CC, Chen SY, Tsai CL, Wu SC, Chiang WC, Wang JL, Sun HY, Chen SC, Chen WJ, Hsueh PR. Prognostic value of mortality in emergency department sepsis score, procalcitonin, and C-reactive protein in patients with sepsis at the emergency department. Shock. 2008 Mar;29(3):322-7. doi: 10.1097/shk.0b013e31815077ca. PMID 17724429
- [Background] Peters RP, Twisk JW, van Agtmael MA, Groeneveld AB. The role of procalcitonin in a decision tree for prediction of bloodstream infection in febrile patients. Clin Microbiol Infect. 2006 Dec;12(12):1207-13. doi: 10.1111/j.1469-0691.2006.01556.x. PMID 17121627